CLINICAL TRIAL: NCT02963792
Title: Values and Virtues in Medical Practice: Quasi-Experimental Intervention for Burnout Preventions, Professionalism Heightening, and Enhancing Resiliency (BUPHER) in a Hospital Surgical Division
Brief Title: Burnout Preventions, Professionalism Heightening, and Enhancing Resiliency (BUPHER)
Acronym: BUPHER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: michal roll (Other Government)
Collaborators: Association for Children at Risk (Other); Tel Aviv University (Other)
Responsible Party: Sponsor-Investigator, michal roll, Principal of the department of surgery and the unit of surgical oncology, Tel-Aviv Sourasky Medical Center
Organization: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TASMC-16-GL-0426-CTIL
Record Dates: First submitted 2016-09-04; First posted 2016-11-15 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Professional-Patient Relations; Burnout, Professional
Keywords: Professionalism; Burnout prevention; Resiliency; Student education
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Structured group intervention (Experimental): Experimental: Structured group intervention a 'structured' intervention, leaning mostly on tools designed to prevent burnout and promote resilience, including predetermined exercises and topics as discussion goals in each meeting.
  Fidelity will be checked and monitored at the end of each meeting, when facilitators fill out a form that summarizes the content, topics and coping skills acquired in each session.
  Interventions: Other: Preventing Professionals burnout
- Semi-Structured group intervention (Experimental): Experimental: Semi-Structured group intervention a 'semi-structured' intervention, based on tools for developing an emotional discourse, building a supporting team and self reflection.
  The 'semi-structured' intervention offers predetermined contents that are discussed through the stories and needs presented by group members.
  Fidelity will be checked and monitored at the end of each meeting, when facilitators fill out a form that summarizes the content, topics and coping skills acquired in each session.
  Interventions: Other: Preventing Professionals burnout

INTERVENTIONS:
Other: Preventing Professionals burnout
  Other Names: Enhancing professional professional conduct

SUMMARY:
Due to their difficult and stressful work surgeons are under continuous physical and mental stress exposing them to increased risk for burnout and lack of professionalism. The present intervention focuses on providing time and a safe space to debrief and explore personal and group experiences and dilemmas, as well as acquire coping skills related to burnout, communication and professionalism.

ELIGIBILITY:
Inclusion Criteria:

* All physicians (residents and experts) of the Surgical Division at Tel Aviv Sourasky Medical Center.
* All medical students studying at the Sackler Faculty of Medicine, Tel Aviv University, and attending a surgery round at the Surgical Division at Tel Aviv Sourasky Medical Center.
* Patients (and/or family members) in the Surgical Division at Tel Aviv Sourasky Medical Center following their surgery.

Exclusion Criteria:

* The research will not include children and/or judgment-impaired patients;
* population not met by inclusion criteria;
* non-Hebrew speaking patients;
* ventilated patients;
* patients in surgical intensive care;
* patients medically defined as suffering from clouding of conscious or delirium;
* subjects who decided to stop their participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Professionalism Culture Scale | Change (increase) from baseline to short and long term measurements (after one year, 3 years, respectively)
  12 item scale developed by the American Board of Internal Medicine, by (DeLisa, Foye, Jain, Kirshblum, & Christodoulou, 2001
Abbreviated Burnout Scale | Change (decrease) from baseline to short and long term measurements (after one year, 3 years, respectively)
  Nine item scale focused on 3 burnout factors (Iverson, Olekalns & Erwin, 1998)

SECONDARY OUTCOMES:
Adapted Professionalism Mini-Evaluation Scale Exercise scale | Change (increase) from baseline to short and long term measurements (after one year, 3 years, respectively)
  originally included 24 items developed by Cruess, McIlroy, Cruess, Ginsburg, and Steinert (2006). Translated and adapted by the research team, and now include 31 items.
Cynicism in Medicine Questionnaire (CMQ) | Change (decrease) from baseline to short and long term measurements (after one year, 3 years, respectively)
  14 item questionnaire developed by Teserman, Morton, Loo, Worthle & Lamberton, 1996
Moral & Cognitive Courage Scale | Change (increase) from baseline to short and long term measurements (after one year, 3 years, respectively)
  A newly developed questionnaire focused on self efficacy to intervene when a physician acts immorally and actual experience with acting in such cases.
Jefferson Health Professionals Empathy Scale | Change (increase) from baseline to short and long term measurements (after one year, 3 years, respectively)
  20 items questionnaire developed by Hojat, Mangione, Nasca, Cohen, Gonnella, Erdmann & Magee, 2001
The Areas of Work life Scale (AWS) | Change (increase in balance) from baseline to short and long term measurements (after one year, 3 years, respectively)
  29 items questionnaire developed by Leiter & Maslach, 2004 to measure 6 factors related to work load, control, appreciation, community, fairness and values
Professionals Self Care Practices questionnaire | Change (increase) from baseline to short and long term measurements (after one year, 3 years, respectively)
  43 items comprised from two questionnaires focused on different aspects of self care (Teng, Yen & Fetzer & Shananfelt et al., 2005). the combination of these two questionnaires was assessed by Karnieli-Miller & Michael.
Life satisfaction questionnaire | Change (increase) from baseline to short and long term measurements (after one year, 3 years, respectively)
  3 item questionnaire focused on general life satisfaction.
Perceived Stress Scale (PSS) | Change (decrease) from baseline to short and long term measurements (after one year, 3 years, respectively)
  10 item scale focused on perceived stress in the clinics (4 items validated in Ben-Zur & Michael) and 6 items developed by the research team to assess concern and fear from medical mistakes and hierarchy.
Work-Life Balance | Change (increase) from baseline to short and long term measurements (after one year, 3 years, respectively)
  6 item questionnaire developed by Greenhaus & Powell, 2006)
Resilient Coping Questionnaire (RCQ) | Change (increase) from baseline to short and long term measurements (after one year, 3 years, respectively)
  24 items questionnaire developed by Wolmer, Hamiel & Laor (2105)
Specific Life Satisfaction Questionnaire | Change (increase) from baseline to short and long term measurements (after one year, 3 years, respectively)
  12 items questionnaire developed by Karnieli-Miller & Michael to measure satisfaction with different life domains (e.g., relationships, financial etc).
Brief Resilience Scale (BRS) | Change (increase) from baseline to short and long term measurements (after one year, 3 years, respectively)
  6 item questionnaire developed by Smith et al., 2008
Patient Satisfaction questionnaire | Change (increase) from baseline to short and long term measurements (after one year, 3 years, respectively)
  23 items questionnaire focused on patient-physician communication skills and satisfaction from care.
Physician Transcendence Scale (PTS) | Baseline
  A 16 items newly developed questionnaire focused on the physicians' transcendence. Laor, Wolmer & Hamiel
Demographic information questions | Baseline
  questions concerning gender, age, seniority, specialty, country of birth,
Life Events Scale | Baseline
  Assessing life events the individual experienced, such as divorce, a death of a loved one, etc.

IPD SHARING:
Plan to Share IPD: Yes
The participants data will be shared with the research team from the Department of Medical Education, Sackler Faculty of Medicine, Tel Aviv University and Cohen-Harris Resilience Center